CLINICAL TRIAL: NCT00866450
Title: Effects of a Western-type Diet on Colorectal Inflammation, Gut Permeability and Systemic Endotoxemia
Brief Title: Effects of a Western-type Diet on Colorectal Inflammation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SWP-0658
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Inflammation
MeSH Terms: interventions — Calcium; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Western style diet (Active Comparator): high-fat, low-calcium diet
  Interventions: Dietary Supplement: Western style diet (high fat and low in calcium)
- Prudent diet (Active Comparator): low-fat, calcium-sufficient diet
  Interventions: Dietary Supplement: Prudent-style diet (low fat and high in calcium)

INTERVENTIONS:
Dietary Supplement: Western style diet (high fat and low in calcium) — Subjects will be randomized to begin on either a WD or a PD for 30 + 3 days. Once that dietary intervention is complete, subjects will have a four (4) week wash-out period and then will be placed on the other dietary intervention for 30 + 3 days
  Arms: Western style diet
Dietary Supplement: Prudent-style diet (low fat and high in calcium) — Subjects will be randomized to begin on either a WD or a PD for 30 + 3 days. Once that dietary intervention is complete, subjects will have a four (4) week wash-out period and then will be placed on the other dietary intervention for 30 + 3 days
  Arms: Prudent diet

SUMMARY:
This study will look at the inflammatory (changes usually associated with infection/injury to the body) and bowel permeability (bowel's ability to allow contents to enter the body) effects of a Western-style diet (high fat and low in calcium) and a prudent-style diet (low fat and high in calcium) on the colon (large bowel). This study may provide information to prevent colorectal cancer in a high-risk population

DETAILED DESCRIPTION:
Hypothesis: Compared to a prudent-style diet, does a western-style diet increase colorectal inflammation thereby increasing gut permeability and causing increased endotoxins and markers of systemic inflammation.

This is a single blind crossover study. Subjects will be randomized to begin on either a WD or a PD for 30 + 3 days. Once that dietary intervention is complete, subjects will have a four (4) week wash-out period and then will be placed on the other dietary intervention for 30 + 3 days. The following study measures are performed during both the dietary intervention study periods. All the baseline tests will be repeated at the end of each dietary intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or post-menopausal ( 2 years after menopause or stopping HRT)healthy female subjects
* Age between 50 and 72 years
* At increased risk for colorectal cancer (this includes those have had a colorectal adenoma excised, or have a first or second degree relative with colorectal neoplasia).

Exclusion Criteria:

* Personal history of cancer other than non-melanoma skin cancer within the past 10 years
* History of hereditary non-polyposis colon cancer
* Intestinal malabsorption, inflammatory bowel disease
* Prior gastrointestinal surgery other than appendectomy or surgery of the esophagus
* Any excess bleeding or coagulation disorders
* Subjects taking anti-coagulants, sterol-binding resins, NSAIDs other than aspirin, < 600mg per day, other study medications, or other multiple medications that might, in the view of the study physicians, alter colonic function or inflammation
* Total cholesterol greater than 240mg/dl, triglycerides > 600mg, LDL-C > 175
* Subjects with a history of coronary artery disease
* HIV positive subjects
* Subjects taking antibiotics, anti-diabetes, hormone replacement therapy, oral, transplanted or injected contraceptives (thyroid hormone therapy is permitted as long as the subject is euthyroid)
* Currently participating in other clinical studies or completed participation in other clinical studies within the last 30 days

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Inflammation in the rectosigmoid epithelium | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention

SECONDARY OUTCOMES:
Circulating endotoxin levels | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention
Expression profiles of pro- and anti-inflammatory genes in rectosigmoid biopsies | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention
Gut permeability | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention
Inflammatory cytokines in the colorectal mucosa and serum | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention
Luminal and adherent gut microbiota | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention
Fecal calprotectin levels in the stool samples | visit 1, 30 days after the first dietary intervention and 30 days after the second dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Swaroop Pendyala, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States